CLINICAL TRIAL: NCT03658174
Title: Upregulating the Nitric Oxide Pathway To Restore Autonomic Phenotype (UNTRAP). A Double Blind Randomised First "Proof of Concept" Direct Translational Study to Explore the Effects of Dietary Nitrate Supplementation on Autonomic Function in Heart Failure Patients
Brief Title: Upregulating the Nitric Oxide Pathway To Restore Autonomic Phenotype (UNTRAP).
Acronym: UNTRAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: National Institute for Health Research Leicester Biomedical Research Centre, Leicester, UK (Other); Loughborough University (Other); University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0675; Edge ID 108647 (Other: University Hospitals of Leicester NHS Trust)
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure; Arrhythmia
Keywords: Nitrate
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich beetroot juice (Active Comparator): 70mls of concentrated beetroot juice to be taken twice a day. This contains 5-6 mmol of inorganic nitrate.
  Interventions: Dietary Supplement: Nitrate-rich beetroot juice
- Nitrate-free beetroot juice (Placebo Comparator): 70mls of concentrated nitrate-free beetroot juice to be taken twice a day. This is an identical juice from which the nitrate has been removed using a standard anion exchange resin.
  Interventions: Dietary Supplement: Nitrate-free beetroot juice

INTERVENTIONS:
Dietary Supplement: Nitrate-rich beetroot juice — 70mls of concentrated beetroot juice containing approximately 5-6 mmol of inorganic nitrate
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Nitrate-free beetroot juice — 70mls of concentrated beetroot juice that has been nitrate-depleted
  Other Names: placebo
  Arms: Nitrate-free beetroot juice

SUMMARY:
Autonomic nervous system dysfunction is known to be associated with an increased risk of heart rhythm abnormalities and sudden cardiac death (SCD) in patients with chronic heart failure - a condition affecting millions of people worldwide. The nitric oxide pathway has been identified as being involved in mediating the effects of the autonomic nervous system on the heart. Recent studies have shown that dietary nitrates can increase the availability of nitric oxide in the body.

This study hopes to find out if dietary nitrate supplementation can help to improve cardiac and autonomic function in patients with heart failure and autonomic dysfunction and reduce the risk of arrhythmias.

DETAILED DESCRIPTION:
20 participants enrolled at the University Hospitals of Leicester NHS Trust will be invited to take a beetroot juice supplement, which naturally contains a high concentration of nitrates, and a nitrate-free (placebo) beetroot supplement. In a double blind way, participants will be randomised to the order in which they receive the 2 treatments with crossover of the treatments. There will be a washout period between the two treatments.

In order to assess cardiac and autonomic function, and risk of heart rhythm abnormalities, tests will be carried out before and after each treatment period

Hypotheses:

* Nitrate supplementation reverses the autonomic dysfunction seen in Chronic Heart Failure (CHF)
* Markers of prognostic significance for predicting SCD, including QT variability index and cardiac restitution properties (R2I2, PERS), are normalised by nitrate supplementation in patients with CHF.
* Nitrate supplementation results in functional improvement in CHF patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female.
* Diagnosed with chronic heart failure - NYHA II-III
* Reduced heart rate variability
* Left ventricle ejection fraction (LVEF) of ≤40%
* Sinus rhythm on 12 lead ECG
* Must have an adequate understanding of written and spoken English
* Female participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
* Able (in the Investigators opinion) and willing to comply with all study requirements

Non-Invasive Programmed Stimulation (NIPS) Sub-Study Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Patients has a pre-existing ICD device with right ventricular apical lead

Exclusion Criteria:

* Myocardial infarction or coronary revascularization within the last 6 months before study enrolment
* NYHA class IV heart failure symptoms
* Persistent Atrial Fibrillation (AF)/Atrial flutter, or paroxysmal AF with frequent recent episodes of prolonged AF
* Patients taking any other nitrate containing medication or supplement (e.g. Isosorbide mononitrate, GTN)
* Patients taking proton pump inhibitors
* Severe pulmonary disease
* Significant renal impairment (eGFR<15)
* Active cancer with life expectancy < 1year
* Patients with significant diabetic or other autonomic neuropathy
* Current or recent (within the last year) cigarette smokers
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Due to undergo any scheduled elective surgery or other procedures requiring general anaesthesia during the study.
* Participant who is inappropriate for placebo therapy
* Subjects who do not have an adequate understanding of written and spoken English
* Any other significant disease or disorder, which in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV) from baseline | 4 weeks and 8 weeks
  Measure of autonomic function
Change in QT variability index (QTVI) from baseline | 4 weeks and 8 weeks
  Marker of arrhythmia risk
Change in Regional Restitution Instability Index (R2I2) from baseline | 4 weeks and 8 weeks
  Marker of ventricular arrhythmia and sudden cardiac death risk
Change in Peak Electrocardiogram Restitution Slope (PERS) from baseline | 4 weeks and 8 weeks
  Marker of ventricular arrhythmia and sudden cardiac death risk

SECONDARY OUTCOMES:
Change in left ventricular function from baseline | 4 weeks and 8 weeks
  LVEF, volumes and filling pressure (E/e ratio)
Change in peak oxygen uptake (VO2max) on cardiopulmonary exercise test from baseline | 4 weeks and 8 weeks
  Maximum oxygen uptake
Change in total exercise time on cardiopulmonary exercise test from baseline | 4 weeks and 8 weeks
  Time to exhaustion on exercise test
Change in the total score on the Minnesota Living With Heart Failure Quality of Life Questionnaire from baseline | 4 weeks and 8 weeks
  Measured using Minnesota Living With Heart Failure Quality of Life Questionnaire, with total score ranging from 0 to 105
Participant compliance with dietary supplement | 4 weeks and 8 weeks
  Compliance as measured using supplement and food diary
Correlation between Non-Invasive Programmed Stimulation (NIPS) derived and exercise ECG derived R2I2 and PERS values | 4 weeks
  Assessment of the correlation between R2I2 and PERS values recorded using NIPS and exercise ECG

CONTACTS AND LOCATIONS:
Overall Officials: Andre Ng, MBChB, PhD, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided